CLINICAL TRIAL: NCT04275895
Title: Interdependency Between Cognitive and Postural Activities in Prematurely Born Children
Brief Title: Cognitive and Postural Activities of Prematurely Born Children
Acronym: COGNIPOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor ; principal investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2019-A02385-52
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Attention Deficit; Mobility; Postural Activity
Keywords: Prematurely born children; Attention function; Posture; Mobility
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Attention performance of a group of prematurely born children will be compared on a classical school chair and a mobile school chair. The same comparison will be made for a group of term born children.
  The perception of the Vertical gravity of the two groups will be evaluated in sitting position, lying to the right side and lying the left side.
  The postural control of the two groups will be evaluated standing on a force plate in three conditions : eyes opened watching a cartoon, eyes opened gazing a fixation cross on the wall and eyes closed.
  The postural control of the two groups will be measured during the execution of three different attentional tasks. For each task, two levels of difficulty will be tested.
  Finally, growth trajectory from birth will be analysed as a confounding factor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prematurely born Children (Experimental): Evaluation of different attention or/and postural activities :
  1. Speed and accuracy answer to visual fish (target) appearance evaluated in two conditions of chair (mobile or classic).
  2. Child perception of the vertical compared to the real vertical
  3. Evaluation of the posture of the child during different visual conditions
  4. Evaluation of the posture of the child during different attention tasks at different levels of difficulty
  Interventions: Behavioral: Evaluation of different attention or/and postural activities
- Term born Children (Active Comparator): Evaluation of different attention or/and postural activities
  1. Speed and accuracy answer to visual fish (target) appearance evaluated in two conditions of chair (mobile or classic).
  2. Child perception of the vertical compared to the real vertical
  3. Evaluation of the posture of the child during different visual conditions
  4. Evaluation of the posture of the child during different attention tasks at different levels of difficulty
  Interventions: Behavioral: Evaluation of different attention or/and postural activities

INTERVENTIONS:
Behavioral: Evaluation of different attention or/and postural activities — 1. The children, equipped with a head-mounted display (HMD), will indicate as quickly as possible the direction of a fish that can be surrounded by congruent or not flankers (Inhibition) and/or preceded by signal (Alert)
  2. The children, equipped with a HMD and a joystick, will vertically turn a randomly inclined stick
  3. The children will stand on a force plate watching a cartoon, gazing a fixation cross or eyes closed
  4. The children, equipped with an augmented reality headset, will perform 2 levels of difficulty of 3 attention tasks standing on a force plate:
     * They will click as quickly as possible when they see a frog among successively appearing animals (vigilance task)
     * They will give the name of an animal appearing at one of the windows displayed (visual search task)
     * They will count the number of yellow lions oriented to the right among several animals of different color and direction (inhibition task)
  5. Growth trajectory will be retrieved from health booklet

SUMMARY:
Prematurely born children (PC) have academic difficulties related to poorer attention capabilities. Additionally, they often show excessive mobility, quoted as agitation. Some consider it could be related to poorer postural control and impaired perception of gravity vertical. But, this excessive mobility could also be an unconscious way for PC to improve their attention performance. The aim of this study is to evaluate the interdependence between postural and cognitive activities in school age PC versus term born children (TC). First, the performance of PC and TC at the Attention Network Test for Children will be analyzed with the use of a mobile versus a classic school chair. Secondly, participants will have to position a stick vertically to measure their perception of vertical gravity. Finally, the spontaneous postural activity of PC and TC (evaluated by the center of pressure displacement) will be studied during the execution of three different attention tasks at different levels of difficulty. Success rate and reaction time will be analyzed for all attention tasks. Moreover, center of pressure displacement calculation will allow evaluation of infants' spontaneous mobility, the precision of their postural control and the attention allocated to their posture.

DETAILED DESCRIPTION:
Prematurely born children (PC) at school age have academic difficulties related to poorer attention capabilities. Posner (1990) described three distinct attention functions: Alert (to maintain a vigilance state), Orientation (to select the relevant information) and Inhibition (to resist distraction). Additionally, teachers and parents are often concerned because they move more than term born children; this excessive mobility being often quoted as agitation. Some consider it would be related to a poorer postural control potentially explained by a poorer perception of vertical gravity. Another explanation is that this mobility could be an unconscious way for PC to increase their arousal level to improve their attention performance. Therefore, the aim of this study is to evaluate the interdependence between postural and cognitive activities in school age PC and term born children (TC). First, the performance of PC and TC at the Attention Network Test for Children will be analyzed evaluating Alert and Inhibition, and its evolution when the infants will use a mobile school chair, compared to a classic school chair. Secondly, participants will perform a test of perception of vertical gravity in which they will have to position a stick vertically. Finally, the spontaneous postural activity of PC and TC (evaluated by the center of pressure displacement measured with a forced plate) will be studied during the execution of three different attention tasks: a vigilance task, a visual search task or an inhibition task at two different levels of difficulty. Success rate and reaction time will be analyzed for all attention tasks. Moreover, center of pressure displacement calculation will allow evaluation of infants' spontaneous mobility, the precision of their postural control and the attention allocated to their posture. Success rate and reaction time will be analyzed for all the attention tasks as well as the angle errors in degree between the stick orientation given by the children and the real vertical. Furthermore, the sway path, the surface area and the entropy of the displacement of CP will be computed to determine respectively the mobility, the precision of the postural control and the attention allocated to the posture of these children.

ELIGIBILITY:
Inclusion Criteria:

* Children born before 37 weeks gestation or at term and routinely followed for their prematurity in the follow-up clinic of the Maternite Regionale Universitaire and healthy term born children recruited after information in different schools of Meurthe-et-Moselle
* Child whose holders of parental authority have received complete information on the organization of the research and have signed the consent

Exclusion Criteria:

* Severe hypotrophy at birth defined by a weight z-score below -2.
* Children with developmental, cognitive, visual or motor disability preventing the execution of the tests

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Accuracy and Reaction time (in msec) to the response to visual target (fish) direction | 8 minutes
  40 trials of fishes displayed for a maximum of 2500 msec to the left or the right hand side, by chair condition (classic, mobile), where the child has to give as quickly as possible the direction of the fish
Angle error (in degree) between the stick orientation given by the child and the real vertical | 4 minutes 30 secondes
  3 trials of randomly inclined stick by position (sitting, lying to the right, lying to the left) where the child has to turn the stick vertically
Sway path (distance traveled by the center of pressure - CP -) and surface area (ellipse covering 90% of the center of pressure displacement) | 4 minutes 30 secondes
  3 x 30 secondes of record on the force plate by standing condition (eyes opened watching a cartoon, gazing a fixation cross, eyes closed) where the child has to stay up without move their feet
Sway path (distance traveled by the center of pressure - CP -), surface area (ellipse covering 90% of the center of pressure displacement) and entropy (index of regularity of postural oscillations) | 12 minutes
  2 x 1 minutes of record on the force plate by level of difficulty (easy, difficult) and by task (vigilance task, visual search task, inhibition task)

CONTACTS AND LOCATIONS:
Locations (1):
- Maternite Regionale Universitaire CHRU NANCY, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No